CLINICAL TRIAL: NCT05894993
Title: Transient Elastograghy to Detect NAFLD in RTRs
Brief Title: Transient Elastograghy to Detect Non Alcoholic Fatty Liver Disease in Renal Transplantation Recipients.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Amany Khaled Ali Ahmed (Other)
Responsible Party: Sponsor-Investigator, Amany Khaled Ali Ahmed, Director, Assiut University
Organization: Assiut University (Other)
Other Study IDs: NAFLD in RTRs
Record Dates: First submitted 2023-05-14; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Renal Transplant Complication Pre-Existing Disease
Keywords: Transient Elastograghy
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: transient elastograghy — is a non-invasive method proposed for the assessment of hepatic fibrosis in patients with chronic liver disease by measuring liver stiffness. It can be easily performed at the bedside or in the outpatients clinic with immediate results and good reproducibility.

SUMMARY:
a. Primary (main): The presence of non alcoholic fatty liver disease in post renal transplantation recipients by non invasive methods as transient elastograghy b-Secondary (subsidiary): to evaluate if transient elastograghy could be used as a noninvasive tool as new perspective on the prediction, prevention of non alcoholic fatty liver disease in renal trasplantation recipients .

DETAILED DESCRIPTION:
. Nonalcoholic fatty liver disease is caused by an accumulation of fat in the liver in the absence of significant alcohol intake. Nonalcoholic fatty liver disease is the most common chronic liver disorder. Chronic kidney disease defined as decreased kidney function shown by glomerular filtration rate (GFR) of less than 60 mL/min per 1•73 m2, or markers of kidney damage, or both, of at least 3 months duration, regardless of the underlying cause.

Nonalcoholic fatty liver disease (and chronic kidney disease constitute a global public health problem, affecting approximately 25% and 10% of the world population, respectively. In recent years, both Nonalcoholic fatty liver disease and chronic kidney disease have shown increasing incidences.

Renal transplantation has significantly improved the survival of patients with end-stage renal disease (ESRD). Despite major advancements in immunosuppressive treatment of renal transplant recipients (RTR) that significantly increased graft and patient short-term survival and lowered the incidence of rejection crises, long-term prognosis is still poor. ., Immunosuppressive drugs used in renal trasplantation increase incidence and severity of traditional cardiovascular risk factors and thus have expected effects on components of the metabolic syndrome (MS) after kidney transplantation. Other Common factors underlying the pathogenesis of and chronic allograft dysfunction may be insulin resistance, oxidative stress, activation of rennin-angiotensin system , Dyslipidemia, and inappropriate secretion of inflammatory cytokines by stereogenic and inflamed liver.

NAFLD represents a liver manifestation of metabolic syndrome and it development is strongly associated with all components of MS in general population. They propose that the presence of NAFLD in RTR could be a strong predictor in cardiovascular morbidity and mortality., Wang H, Lin ZT, Yuan Y, Wu T. hypothesis that non alcoholic fatty liver disease may be associated with deteriorating graft function, causing a chronic allograft nephropathy and graft loss.

Due to the high rate of corticosteroid askwith considering the strong relationship between chronic kidney disease and NAFLD, NAFLD would probably be a common disorder among kidney transplantation recipients if these patients did not receive stereogenic medications.

ELIGIBILITY:
Inclusion Criteria:

* • a. Inclusion criteria: All renal transplant recipients with a functioning graft for more than 1 year coming for follow up at renal outpatient clinics in Assiut university hospitals .

  * Trough level of immunosuppressive drugs .

Exclusion Criteria:

* Patients are excluded for participation in the study if

  * chronic hepatitis B and/or C virus infection,
  * CMV infections
  * Chronic liver disease
  * presence of other autoimmune or cholestatic liver disease,
  * drug induced liver disorder
  * excessive alcohol abuse,
  * pregnancy
  * malignancy
  * dyslipidemia, bleeding tendency ,
  * Renal rejections .

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All renal transplant recipients with a functioning graft for more than 1 year coming for follow up at renal outpatient clinics in Assiut university hospitals .
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
): The presence of NAFLD in post renal transplantation recipients by non invasive methods as transient elastograghy. | Degree of hepatic fibroses from f0-f4,Degree of steatosis "through study completion, an average of 1 year"
  ): to evaluate if transient elastograghy could be used as a noninvasive tool as new perspective on the prediction, prevention of non alcoholic fatty liver desease in renal trasplantation recipients .

REFERENCES:
- [Result] Gahm C, Park S. The association between skipping breakfast and chronic kidney disease. Int Urol Nephrol. 2023 Dec;55(12):3209-3215. doi: 10.1007/s11255-023-03590-5. Epub 2023 Apr 24. PMID 37093440